CLINICAL TRIAL: NCT05137210
Title: Identifying Efficient Linkage Strategies for Men
Acronym: IDEaL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Partners in Hope, Inc. (Industry); Boston University (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Charles University, Czech Republic (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Kathryn L. Dovel, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INV-001423; INV-001423 (Other: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2021-05-28; First posted 2021-11-30 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hiv
Keywords: HIV self-testing (HIVST); HIV; Antiretroviral therapy (ART); ART Initiation; ART Retention; Men; HIVST
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Male-specific counseling and facility navigation (Experimental)
  Interventions: Other: Male Counseling and Facility Navigation
- Home-Based ART Initiation (Experimental)
  Interventions: Other: Home-Based ART Initiation and Facility Navigation
- Stepped Intervention (Experimental)
  Interventions: Other: Stepped Intervention

INTERVENTIONS:
Other: Male Counseling and Facility Navigation — At enrollment, study staff distribute pamphlet with male-specific messaging and contact information for nearest facility. Low-level cadre traces participants and provides one-on-one, in person male-specific counseling. Meeting at location of participants choice. Follow-up male-specific counseling is offered every 14 days thereafter until 90 days is reached OR 4-week follow-up ART refill visit is completed. Participants who choose to initiate ART are escorted to nearest health facility and provided facility navigation assistance.
  Arms: Male-specific counseling and facility navigation
Other: Home-Based ART Initiation and Facility Navigation — At enrollment, study staff distribute two pamphlets on: 1) male-specific messaging and 2) details about home-based ART initiation. Low-level cadre traces participants and provides one-on-one, in person male-specific counseling, and a detailed description of home-based ART initiation with a nurse. Meeting at the location of participants choice. Follow-up male-specific counseling and information about home-based initiation is offered every 14 days thereafter until 90 days OR 4-week ART follow-up refill visit is complete. Participants who choose to initiate ART at home or in the community will meet with a nurse at a place of the participants choosing. Those who choose to initiate at the facility will receive facility navigation and initiation. All clients will receive a "warm handover" for their 4-week ART follow-up visit.
  Arms: Home-Based ART Initiation
Other: Stepped Intervention — Day 0-14 Arm 1 (Male-specific counseling and facility navigation arm) implemented. Day 14-30, if not yet initiated, a psychosocial counsellor will trace the participant to provide advanced counselling and motivational interviewing. Psychosocial counsellors will act as 'Male Mentors' and meet with men as frequently as needed. Day 30-89 if not yet initiated, nurse-led home-based ART initiation will be offered, following the same steps as listed in the "Home-Based ART Initiation" Arm.
  Arms: Stepped Intervention

SUMMARY:
HIV self-testing (HIVST) has been found to be a highly acceptable approach for men to learn of their HIV status and has resulted in increased testing uptake. However, rates of antiretroviral therapy (ART) initiation among those tested with HIVST are difficult to capture. This clinical trial will test varying approaches to ART initiation and retention among men who test positive using HIVST to learn about the most effective strategy to engage men in ART services.

DETAILED DESCRIPTION:
HIV self-testing (HIVST) has been found to be a highly acceptable approach for men to learn of their HIV status and has resulted in increased testing uptake. However, rates of antiretroviral therapy (ART) initiation among those tested with HIVST are difficult to capture and some studies have suggested that linkage rates are low , particularly amongst men. The investigators propose a clinical trial to test varying approaches to ART initiation and retention among men who test HIV-positive through HIVST. Three interventions will be tested:

Standard of Care (Arm 1): phone and in-person follow-up, accompanied with male-specific counseling (given every two weeks for up to 90-days or until ART initiation is achieved, whichever comes first); Home-Based ART initiation (Arm 2): nurse-led ART initiation at home or in the community Staged Intervention (Arm 3): a staged intervention that consecutively increases in intensity every month that a participant does not initiate ART (intervals include: Days 1-14: Standard of Care; Days 14-30: Peer support with a psychosocial consellor; Days 30-90: Nurse-led Home-Based ART initiation);

The primary objective is to identify a cost-effective package comprised of male-specific counseling, peer support, community ART distribution and/or home-based ART services for ART initiation and retention among men identified as HIV-positive through HIVST in Malawi. The specific objectives are:

Aim 1. Evaluate the effectiveness of the Stepped ART Intervention (Arm 3) vs male counseling and facility navigation (Arm 1) (primary analysis) and the effectiveness of the Stepped ART Intervention (Arm 3) vs home-based ART initiation with a nurse (Arm 2) (secondary analysis) on ART initiation within 4-months after enrollment in the trial.

Aim 2. Identify individual-, community-, and facility-level factors associated with ART initiation within each intervention arm (male counseling, home-based ART and Stepped intervention) using baseline and semi-structured in-depth interviews.

Aim 3. Determine the cost-effectiveness and scalability of the intervention arms through costing and mathematical modeling.

An individually randomized control trial will be performed with 545 HIV-positive men. Men will be individually randomized 1:1:1 to one of the three intervention arms described above. They will receive their assigned intervention over the course of three months or until the participant initiates ART. The study will be preformed at 10 health facilities supported by Partners in Hope (PIH). Data collection will include baseline and follow-up surveys at 2- and 4-months; medical charter reviews at 2- and 4-months after study enrollment; qualitative interviews with a subset of men and their female partners; and a cost analysis of costs associated with each arm. Male participants will be enrolled in the study for a total of 4 months.

The investigators anticipate learning about the most effective stragty to engage men in ART. The investigators also anticipate learning about the type and degree of followup necessary to support men's engagement in ART services. Finally, the investigators anticipate learning about the cost-effectiveness of intervention, with the goal of improving cost-effectiveness for the Ministry of Health. Results from this study could be used to define best practices and to further scale ART-focused programs for men in Malawi.

ELIGIBILITY:
Men:

Inclusion Criteria:

* ≥15 years of age
* Tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Not currently engaged in ART services, defined as:

  * Tested HIV-positive ≥14 days and not on ART ≥14 days after testing HIV-positive;
  * ≥14 days late for the first four-week follow up appointment; or
  * Initiated ART but ≥60 days late for last ART appointment;
  * Has not taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living inside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Exclusion Criteria:

* <15 years of age
* Never tested HIV positive using Ministry of Health standard algorithm (Determine + Unigold)
* Tested HIV-positive <14 days ago
* Currently engaged in ART services, defined as:

  * Initiated ART
  * <14 days late for the first four-week follow up appointment
  * Initiated ART and <60 days late for last ART appointment
  * Has taken ART in the past 7-days, as indicated by a point of care (POC) urine assay
  * Living outside the facility catchment area (defined as any area that HCWs from the study facility routinely visit for tracing purposes)

Female partner

Inclusion Criteria:

* ≥15 years of age
* Male partner enrolled in the study
* Male partner agrees that the female can be recruited for an in-depth interview

Exclusion Criteria:

* <15 years of age
* Male partner is not enrolled in the study
* Male partner does not agree that the female can be recruited for an in-depth interview

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 569 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of men who are retained on ART early | 4-months.
  Proportion of men who initiate ART at 3-months and attended their 4-week ART refill appointment at 4-month after enrollment. Sourced from medical chart reviews.

SECONDARY OUTCOMES:
Proportion of men who initiate ART | 3-months
  Proportion of men who initiate at 3-months after enrollment. Sourced from medical chart reviews.
Any adverse events self-reported by female ART client or male partner | 4-months
  Self-report of any adverse event from female ART client (IPV, unwanted disclosure, end of relationship) and their male partners (unwanted disclosure) who were identified as HIV-positive. Sourced from follow-up surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners in Hope, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in an article after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning three months and ending five years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be sent to Dr. Dovel (kdovel@mednet.ucla.edu). To gain access, data requestors will need to sign a data access agreement. Data are available for five years.

REFERENCES:
- [Derived] Hubbard J, Mphande M, Robson I, Balakasi K, Phiri K, Chikuse E, Thorp M, Phiri S, Choko AT, Cornell M, Coates T, Dovel K. Core components of male-specific person-centred HIV care: a qualitative analysis from client and healthcare worker perspectives in Malawi. BMJ Public Health. 2024 Dec 22;2(2):e001100. doi: 10.1136/bmjph-2024-001100. eCollection 2024 Dec. PMID 40018627
- [Derived] Holland KN, Hubbard J, Mphande M, Robson I, Phiri K, Onoya D, Chikuse E, Dovel K, Choko A. Implementation of Male-Specific Motivational Interviewing in Malawi: An Assessment of Intervention Fidelity and Barriers to Scale-Up. medRxiv [Preprint]. 2024 Sep 26:2024.09.24.24314326. doi: 10.1101/2024.09.24.24314326. PMID 39399024
- [Derived] Dovel K, Balakasi K, Hubbard J, Phiri K, Nichols BE, Coates TJ, Kulich M, Chikuse E, Phiri S, Long LC, Hoffman RM, Choko AT. Identifying efficient linkage strategies for men (IDEaL): a study protocol for an individually randomised control trial. BMJ Open. 2023 Jul 12;13(7):e070896. doi: 10.1136/bmjopen-2022-070896. PMID 37438067